CLINICAL TRIAL: NCT07084103
Title: Effectiveness of a Psychosocial Support Intervention for Women Diagnosed With Fetal Anomaly: Randomised Controlled Trial
Brief Title: Effectiveness of a Psychosocial Support Intervention for Women Diagnosed With Fetal Anomaly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-16214662-050.01.04-305615
Record Dates: First submitted 2025-06-30; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Fetal Diseases; Congenital Abnormalities; Pregnant Women; Psychosocial Support Systems; Mental Health
Keywords: Fetal anomaly; Congenital abnormalities; Psychosocial support; Psychological intervention; Pregnant women; Prenatal diagnosis; Mental health; Coping strategies; Emotional well-being
MeSH Terms: conditions — Fetal Diseases; Congenital Abnormalities; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants in the control arm will receive routine prenatal care as provided by their healthcare providers. No additional psychosocial support or structured intervention will be administered beyond the standard medical and obstetric services.
- "Psychosocial Support Intervention" (Experimental): Participants in the intervention arm will receive a structured psychosocial support program designed for women diagnosed with fetal anomaly. The program includes individual counseling sessions, stress management techniques, emotional support, and educational materials addressing coping strategies and mental well-being. The intervention will be delivered by trained healthcare professionals over sessions during the prenatal period.
  Interventions: Behavioral: Psychosocial Support Intervention

INTERVENTIONS:
Behavioral: Psychosocial Support Intervention — Participants in the intervention arm will receive a structured psychosocial support program designed for women diagnosed with fetal anomaly. The program includes individual counseling sessions, stress management techniques, emotional support, and educational materials addressing coping strategies and mental well-being. The intervention will be delivered by trained healthcare professionals over sessions during the prenatal period.
  Arms: "Psychosocial Support Intervention"

SUMMARY:
This study aims to evaluate the effectiveness of a psychosocial support intervention for women diagnosed with fetal anomaly. A randomized controlled trial design will be used, and women diagnosed with fetal anomaly will be included as participants. The intervention group will receive a structured psychosocial support program, while the control group will receive routine care.

DETAILED DESCRIPTION:
Providing psychosocial support to pregnant women to maintain their psychosocial health plays a facilitating role in helping them acquire the knowledge and skills necessary to cope with the difficulties they encounter, facilitating their functional adaptation and improving their quality of life. In the presence of a foetus with a diagnosis of anomaly risk during pregnancy, it becomes even more important for pregnant women to receive psychosocial support to protect their mental and physical health.

The main objective of this project is to examine the effectiveness of online psychosocial support provided to pregnant women with foetuses at risk of anomaly during their pregnancy. In line with this main objective, the psychosocial support needs of pregnant women with a risk of foetal abnormalities will first be determined using a qualitative research design. Subsequently, the effectiveness of the online psychosocial support developed in line with these needs will be objectively demonstrated in pregnant women with a risk of foetal abnormalities using a randomised controlled research design and measurement tools.

ELIGIBILITY:
Inclusion Criteria:

* In her current pregnancy, the results of the dual or triple screening test (a screening test result of 1:50 or 1:100 is considered a high risk for Down syndrome (Şirin, 2020) and/or ultrasound findings (physical/anatomical and congenital anomalies) indicate a high risk of foetal abnormalities,
* Decision to continue the pregnancy,
* Being over 18 years of age,
* Having received hospital services at least once after the initial diagnosis (this criterion was added to enable the pregnant woman to evaluate the services she received from the hospital after the diagnosis and to express her expectations beyond the services provided)
* No mental or psychological disorders that would make it difficult to express oneself,
* Voluntary participation in the study.

Exclusion Criteria:

• Pregnant women who do not meet the inclusion criteria will be excluded from the sample.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Level of depression, anxiety and stress | Pre-test data: before the 20th week of pregnancy Post-test data: after a 6-week intervention Follow-up data: 4 weeks after the post-test Second follow-up data: 6 weeks after the birth
  It will be measured using the "Depression-Anxiety-Stress Scale". This scale is a 4-point Likert-type scale with responses ranging from '0 = never' to '3 = always' and consists of seven questions measuring 'depression, stress and anxiety dimensions'.
Level of prenatal attachment | Pre-test data: before the 20th week of pregnancy Post-test data: after a 6-week intervention Follow-up data: 4 weeks after the post-test
  It will be measured using the "Prenatal Attachment Inventory". The scale, which consists of 21 items, was developed to describe the thoughts, feelings, and situations experienced by women during pregnancy and to determine their level of attachment to their baby during the prenatal period. Each item is scored on a four-point Likert scale ranging from 1 to 4. A score of at least 21 and a maximum of 84 can be obtained from the scale. An increase in the score obtained by the pregnant woman indicates an increase in the level of attachment. The items are scored as follows: 1: Never, 2: Sometimes, 3: Often, 4: Always.
Level of maternal attachment | 6 weeks after the birth
  "The Maternal Attachment Scale" will be used to measure maternal attachment. Each item is a 26-item, four-point Likert-type scale ranging from 'always' to 'never.' Each item contains direct statements and is scored as follows: Always = 4, Often = 3, Sometimes = 2, and Never = 1. A total score is obtained from the sum of all items. A high score indicates a high level of maternal attachment. The lowest possible score from the scale is 26, and the highest is 104. A high score on the scale indicates a high level of maternal attachment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Türkiye/Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol